CLINICAL TRIAL: NCT01040481
Title: Laparoscopic Revisional Surgery: Adding Malabsorption for Failed Gastric Bypass
Brief Title: Adding Malabsorption for Failed Gastric Bypass
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD, FACS; FASMBS; Professor of Surgery, University of California San Francisco, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2009066; U1111-1113-0500 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-26; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Clinically Severe Obesity; Obesity Recidivism; Inadequate Initial Weight Loss; Poor Weight Loss; Persistent Obesity; Refractory Obesity; Intractable Obesity
Keywords: Failed gastric bypass; Malabsorptive distal gastric bypass; Distal gastric bypass; Malabsorptive gastric bypass; Adding malabsorption; Increasing malabsorption; Re-operative bariatric surgery; Revisional bariatric surgery; Revisional gastric bypass; Reoperations; Conversions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Malabsorptive distal gastric bypass

SUMMARY:
The main aim of this study is to analyze and report the preliminary and intermediate term outcomes after laparoscopic revision Roux-en-Y gastric bypass surgery for weight recidivism. The foremost outcome measurements are 1) Fat loss mainly measured as weight loss and expressed as trends in BMI, %EWL, and/or %EBL; 2) Trend in Comorbidity status; and 3) Patient satisfaction and Health-Related Quality of Life "HR-QoL" measured by a standardized, non-validated subjective satisfaction questionnaire and the validated, disease-specific, Moorehead-Ardelt II QoL questionnaires, respectively; 4) Morbidity & Mortality including nutritional status and metabolic complications.

Consequently, secondary objectives of this study are 1) to assess failure rate defined as percentage of excess weight loss < 50% , lowest BMI >35 for morbidly obese (MO) or >40 for superobese (SO), and/or lack of resolution/improvement of major comorbidities at the point in time when assessing preliminary and intermediate results after the surgery under analysis. 2) To evaluate the metabolic and nutritional status by measurements of particular clinical and biochemical parameters.

This research is in line with the most current provocative new ideas and recent high impact publications. To the best of our knowledge, this is the very first outcome study of revisional malabsorptive distal gastric bypass surgery by laparoscopy with diverse revisional strategies such as revisional gastroplasty, revisional Fobi-Capella, revisional Adjustable Gastric Band, conversion to distal, and conversion to very, very long limb gastric bypass. Previously, several studies have addressed conversion to malabsorptive gastric bypass after a failed primary proximal gastric bypass but none has addressed the failed distal gastric bypass nor the adequate balance between increasing restriction and malabsorption for decreasing the risk of protein-calorie malnutrition.

DETAILED DESCRIPTION:
Since 1998, there has been a substantially progressive increase in bariatric surgery. In 2005, the American Society of Metabolic and Bariatric Surgery (ASMBS) reported that 81% of bariatric procedures were approached laparoscopically. 205,000 people, in 2007, had bariatric surgery in the United States from which approximately 80% of these were Gastric Bypass. Moreover, there is a mismatch between eligibility and receipt of bariatric surgery with just less than 1% of the eligible population being treated for morbid obesity through bariatric surgery. Along with the increasing number of elective primary weight loss procedures, up to 20% of post RYGB patients cannot sustain their weight loss beyond 2 to 3 years after the primary bariatric procedure11. Thus, revisional surgery for poor weight loss and re-operations for technical or mechanical complications will rise in a parallel manner. RYGB is consistently considered the revisional procedure of choice for failed restrictive procedures.

At present there are three broad categories of bariatric procedures according to its mechanism of action: 1) purely restrictive, 2) primarily restrictive with some malabsorption, and 3) primarily malabsorptive with some restriction. Modern standard bariatric procedures recognized by the American Society for Metabolic and Bariatric Surgery "ASMBS" include the following 1) adjustable gastric band, 2) sleeve gastrectomy, 3) gastric bypass, 4) biliopancreatic diversion, and 5) duodenal switch.

In general, there is a lack of long-term (5-10 years) and very long-term (> 10 years) outcome studies for modern bariatric surgery that would allow us to better define the role of each one of these procedures, especially after the advent of the laparoscopic approach.

In an animal model, diet induced obese animals exhibiting metabolic syndrome underwent Roux-en-Y gastric bypass with highly reproducible surgical outcomes as well as biochemical and energetic homeostatic abnormalities similar to post-RYGB findings in humans. Weight regain occurs in approximately 20% of patients after two to three years after RYGB. It seems that the weight-loss-promoting effects of chronically elevated plasma PYY concentrations dominate the weight-gain-promoting effects of lowered plasma leptin concentrations, with the relative plasma PYY: leptin concentration ratio determining whether weight loss will be sustained or regained.

Several studies have compared different Roux limb lengths in primary bariatric surgery. It seems to be that long limb RYGB (150cm), especially in patients with BMI > 50 kg/m2, confers at least better short-term weight loss without nutritional consequences. Conversely, other investigators have not found any clinically significant difference in weight loss with increasing Roux limb lengths, especially in patients with BMI < 50 kg/m2 23-26. The following are the main investigators that have increased the malabsorptive component of the failed proximal gastric bypass as a revisional strategy:

1. Torres JC in 1991 was the first to propose this strategy with a cohort of 140 patients followed for 5 years (90.5% follow-up rate). Analyzed traditional outcome measures were early (2.1%) and late (27%) morbidity including protein-calorie malnutrition (7%); %EWL at 1,2,3,4,and 5 years were 89.5%, 91%, 87%, 82.5%, 82.5%, respectively; and re-operations.
2. Fox SR and Oh KH et al in 1996 reported 10 failed proximal gastric bypass patients undergoing distal gastric bypass from an diverse group of failed primary surgeries (n=80) followed for 3 years with a 92.5% follow-up rate. Reported traditional outcome measures were early (39%) and late (84%) morbidity; %EWL at 1,2,&3 years was 83%, 89%and 94%, respectively; high satisfaction was also reported.
3. Sugerman et al in 1997 published their outcomes with 27 patients. Five patients were converted to a malabsortive distal gastric bypass with a 50cm common channel which required a second revision for malnutrition and two died. 22 patients were revised to a 150cm common channel; three patients required a second revision for malnutrition but %EWL went from 30% to 61% at 1 year and 69% at 5 years. They concluded that a 50cm common channel had an unacceptable morbidity and mortality.
4. Fobi et al in 2000 presented his results of 65 patients after mostly failed primary Fobi pouch operation. 15 patients developed protein calorie malnutrition requiring supplemental nutrition and 6 required further revision.
5. The 2001 Sapala´s et al partial outcome analysis on 303 varied revisionary micropouch gastric bypass procedures with a 200cm Roux limb, 150cm biliopancreatic limb and >200cm common channel. %EWL during 3 years is similar to the primary procedure (68.6%, 76.6%, and 72.3%). However no subset analysis is performed.
6. Pareja et al analysis of 41 patients, undergoing diverse distal malabsorptive techniques, included 32 revisionary procedures after primary Fobi-Capella gastric bypass. At 11, 16, and 19 months of mean follow-up, %EWL for the Scopinaro-style, Brolin, and Fobi revisionary gastric bypasses were 69.7%, 65.0%, 74.8%, respectively. Failure and success rates according to Biron et al. are provided but no other subgroup analysis is provided.
7. Brolin et al on 2007 reported 47 out of 54 patients undergoing revision for failed primary bariatric surgery had a very, very long limb gastric bypass with a 75cm to 100cm common channel and a 15cm to 25cm biliopancreatic limb. 7.4% (n=4) developed protein-calorie malnutrition from which one required 6 weeks of TPN, two elongation of the common channel (150cm) and one reversal after a prolonged hiatus returning with severe metabolic complications. 47.9% of the series lost at least 50% EWL at 1 year. There was no difference between those with primary failed restrictive vs. primary failed gastric bypass patients.
8. Sarr et al on 2007 states that "patients with anatomically intact, non-malabsorptive RYGB when converted to a malabsortive distal RYGB, good results are not common".

To the best of our knowledge and after extensive literature search, there is no outcome study employing a laparoscopic approach for revisional malabsorptive distal Roux-en-Y gastric bypass specially increasing the restrictive component in a failed primary malabsorptive distal type of gastric bypass. Thus, we decided to analyze our own series including the learning curve and diverse revisional techniques in this unique subset of patients: 1) revision gastroplasty; 2) Fobi-Capella (static band); 3) Adjustable gastric band; 4) Conversion to either modality of malabsorptive distal gastric bypass, very, very long limb or distal.

Summarizing, there is lack of very-long term outcomes after bariatric surgery and standardization of gastric bypass surgery. The treatment of inadequate weight loss or weight recidivism after Roux-en-Y gastric bypass (RYGB) remains refractory to medical treatment. Failure rates have been reported up to 20% and 35% for the morbidly obese and super obese, respectively at 2 to 3 years after surgery. The indication for further surgical intervention remains controversial, as does what type of procedure to recommend. Furthermore, there is no standardization of the limb lengths, pouch size or the use of prosthetic reinforcement. Therefore the approach to these patients must be as individualized as their original operations. We analyze our experience with the laparoscopic approach to these complex and challenging patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met NIH criteria for recommendation of a bariatric procedure with the combination of the following characteristics:

  * Failed primary proximal gastric bypass with subsequent revision to a malabsortive distal gastric bypass.
  * Failed primary distal malabsorptive gastric bypass with subsequent revision to increase the restrictive component (revisional: gastroplasty, Fobi, or adjustable gastric band)

Exclusion Criteria:

* Patients with prior major conversions or revisions.
* Missing records and/or unreachable patients with scant information for analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had either clinically severe obesity (morbid obesity, MO, or super obesity, SO) underwent a primary Roux-en-Y gastric bypass. The ones that were subsequently revised ending up with an optimized malabsorptive distal gastric bypass were identified from our prospectively maintained bariatric database and included in this study. Specific metabolic and nutritional complications after RYGB surgery were defined according to standard definitions based on signs, symptoms, and laboratory measurements.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2009-08; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality | throughout follow-up
Weight loss expressed as Body Mass Index and Percentage excess weight loss | throughout follow-up

SECONDARY OUTCOMES:
Traditional outcome measurements | Variable
Remission or improvement of comorbidities | throughout follow-up
Health-related Quality of Life (HR-QoL) | at last follow-up
Subjective Satisfaction | at the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] http://www.asbs.org/htm/Private/resolution.html. American Society for Metabolic and Bariatric Surgeons.
- [Background] O'Brien PE, McPhail T, Chaston TB, Dixon JB. Systematic review of medium-term weight loss after bariatric operations. Obes Surg. 2006 Aug;16(8):1032-40. doi: 10.1381/096089206778026316. PMID 16901357
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Christou NV, Look D, Maclean LD. Weight gain after short- and long-limb gastric bypass in patients followed for longer than 10 years. Ann Surg. 2006 Nov;244(5):734-40. doi: 10.1097/01.sla.0000217592.04061.d5. PMID 17060766
- [Background] Brolin RE. Long limb Roux en Y gastric bypass revisited. Surg Clin North Am. 2005 Aug;85(4):807-17, vii. doi: 10.1016/j.suc.2005.03.003. PMID 16061087
- [Background] MacLean LD, Rhode BM, Nohr CW. Long- or short-limb gastric bypass? J Gastrointest Surg. 2001 Sep-Oct;5(5):525-30. doi: 10.1016/s1091-255x(01)80091-3. PMID 11986004
- [Background] Choban PS, Flancbaum L. The effect of Roux limb lengths on outcome after Roux-en-Y gastric bypass: a prospective, randomized clinical trial. Obes Surg. 2002 Aug;12(4):540-5. doi: 10.1381/096089202762252316. PMID 12194548
- [Background] Lee S, Sahagian KG, Schriver JP. Relationship between varying Roux limb lengths and weight loss in gastric bypass. Curr Surg. 2006 Jul-Aug;63(4):259-63. doi: 10.1016/j.cursur.2006.05.001. PMID 16843777
- [Background] Ciovica R, Takata M, Vittinghoff E, Lin F, Posselt AM, Rabl C, Stein HJ, Campos GM. The impact of roux limb length on weight loss after gastric bypass. Obes Surg. 2008 Jan;18(1):5-10. doi: 10.1007/s11695-007-9312-y. Epub 2007 Dec 7. PMID 18064526
- [Background] Bruder SJ, Freeman JB, Brazeau-Gravelle P. Lengthening the Roux-Y Limb Increases Weight Loss after Gastric Bypass: a preliminary report. Obes Surg. 1991 Mar;1(1):73-77. doi: 10.1381/096089291765561501. PMID 10715665
- [Background] Freeman JB, Kotlarewsky M, Phoenix C. Weight loss after extended gastric bypass. Obes Surg. 1997 Aug;7(4):337-44. doi: 10.1381/096089297765555593. PMID 9730521
- [Background] Feng JJ, Gagner M, Pomp A, Korgaonkar NM, Jacob BP, Chu CA, Voellinger DC, Quinn T, Herron DM, Inabnet WB. Effect of standard vs extended Roux limb length on weight loss outcomes after laparoscopic Roux-en-Y gastric bypass. Surg Endosc. 2003 Jul;17(7):1055-60. doi: 10.1007/s00464-002-8933-4. Epub 2003 May 6. PMID 12728380
- [Background] Inabnet WB, Quinn T, Gagner M, Urban M, Pomp A. Laparoscopic Roux-en-Y gastric bypass in patients with BMI <50: a prospective randomized trial comparing short and long limb lengths. Obes Surg. 2005 Jan;15(1):51-7. doi: 10.1381/0960892052993468. PMID 15760498
- [Background] Torres JC. Why I Prefer Gastric Bypass Distal Roux-en-Y Gastroileostomy. Obes Surg. 1991 Jun;1(2):189-194. doi: 10.1381/096089291765561268. PMID 10775917
- [Background] Fox SR, Fox KS, Oh KH. The Gastric Bypass for Failed Bariatric Surgical Procedures. Obes Surg. 1996 Apr;6(2):145-150. doi: 10.1381/096089296765557097. PMID 10729855
- [Background] Sugerman HJ, Kellum JM, DeMaria EJ. Conversion of proximal to distal gastric bypass for failed gastric bypass for superobesity. J Gastrointest Surg. 1997 Nov-Dec;1(6):517-24; discussion 524-6. doi: 10.1016/s1091-255x(97)80067-4. PMID 9834387
- [Background] Fobi MA, Lee H, Igwe D Jr, Felahy B, James E, Stanczyk M, Tambi J, Eyong P. Revision of failed gastric bypass to distal Roux-en-Y gastric bypass: a review of 65 cases. Obes Surg. 2001 Apr;11(2):190-5. doi: 10.1381/096089201321577866. PMID 11355025
- [Background] Sapala JA, Wood MH, Sapala MA, Schuhknecht MP, Flake TM Jr. The micropouch gastric bypass: technical considerations in primary and revisionary operations. Obes Surg. 2001 Feb;11(1):3-17. doi: 10.1381/096089201321454042. PMID 11361165
- [Background] Brolin RE, Cody RP. Adding malabsorption for weight loss failure after gastric bypass. Surg Endosc. 2007 Nov;21(11):1924-6. doi: 10.1007/s00464-007-9542-z. Epub 2007 Sep 3. PMID 17768659
- [Background] Pareja JC, Pilla VF, Callejas-Neto F, Coelho-Neto Jde S, Chaim EA, Magro DO. [Gastric bypass Roux-en-Y gastrojejunostomy--conversion to distal gastrojejunoileostomy for weight loss failure--experience in 41 patients]. Arq Gastroenterol. 2005 Oct-Dec;42(4):196-200. doi: 10.1590/s0004-28032005000400002. Epub 2006 Jan 19. Portuguese. PMID 16444372
- [Background] Sarr MG. Reoperative bariatric surgery. Surg Endosc. 2007 Nov;21(11):1909-13. doi: 10.1007/s00464-007-9536-x. Epub 2007 Aug 19. No abstract available. PMID 17705073
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery/